CLINICAL TRIAL: NCT03560687
Title: CardioSideral Heart Surgery: Randomized Study on Sucrosomial Iron Supplementation
Brief Title: CardioSideral Heart Surgery: Randomized Study on Sucrosomial Iron Supplementation Before Heart Surgery
Acronym: CHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Principal Investigator, Luca Weltert, Clinical Professor, Principal Investigator, Cardiochirurgia E.H.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-1
Record Dates: First submitted 2018-06-07; First posted 2018-06-18 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Anemia
Keywords: Anemia; Heart Surgery; Iron Supplementation
MeSH Terms: conditions — Anemia | interventions — sucrosomial iron

STUDY DESIGN:
Intervention Model Description: Randomization of 1000 consecutive patients undergoing heart surgery to either Iron supplementation or Control
Who Masked: Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CardioSIDERAL (Experimental): Adminsitration of 2 pills per day of CArdiosideral from 30 days before operation to time of operation
  Interventions: Drug: Sucrosomial Iron
- Control (No Intervention)

INTERVENTIONS:
Drug: Sucrosomial Iron — CardioSideral 2 caps per day
  Other Names: CardioSideral
  Arms: CardioSIDERAL

SUMMARY:
This randomized, single blind (Outcomes Assessor), non-profit study is aimed at verifying whether routine preoperative supplementation with Sucrosomial® Iron in patients scheduled for cardiac surgery may increase baseline haemoglobin, constrain the haemoglobin decrease between postoperative day 2 and 3 (haemoglobin drift), and reduce the postoperative transfusion requirements, in order to identify a new strategy for pre-hospitalization optimization and post-operative recovery.

DETAILED DESCRIPTION:
This randomized, single blind (Outcomes Assessor), non-profit study is aimed at verifying whether routine preoperative supplementation with Sucrosomial® Iron in patients scheduled for cardiac surgery may increase baseline haemoglobin, constrain the haemoglobin decrease between postoperative day 2 and 3 (haemoglobin drift), and reduce the postoperative transfusion requirements, in order to identify a new strategy for pre-hospitalization optimization and post-operative recovery.

Secondary Objectives are

* Changes in blood chemistry and biochemical tests between pre- and post-intervention
* Evaluation of tolerability and compliance of supplementation with Sucrosomal Iron
* Reduction in the number of transfusions and blood bags used
* Evaluation of cost-effectiveness

ELIGIBILITY:
Inclusion Criteria:

Undergoing elective Heart Surgery -

Exclusion Criteria:

- Emergent or Urgent Indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1023 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Preoperative Hemoglobin Level | 30 days from enrollment
  Preoperative Hemoglobin Level

SECONDARY OUTCOMES:
Compliance to drug | 30 days from enerollemnt
  Discontinuation rate due to adverse effects
Cost-effectiveness in terms of cost of drug vs saved blood units | 30 days after operation
  Cost-effectiveness in terms of cost of drug vs saved blood units
Hemoglobin Level 24 hours after operation | 24 hours after index operation
  Hemoglobin Level 24 hours after operation
Hemoglobin Level 48 hours after operation | 48 hours after index operation
  Hemoglobin Level 48 hours after operation

CONTACTS AND LOCATIONS:
Overall Officials: Luca Weltert, Principal Investigator — European Hospital
Locations (1):
- Cardiochirurgia European Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weltert LP, De Rosa A, Rondinelli MB, Falco M, Turani F, Pierelli L. Benefits of pre-operative oral Sucrosomial(R) iron supplementation in cardiac surgery: influence of patient's baseline hemoglobin and gender. Blood Transfus. 2023 Jul;21(4):305-313. doi: 10.2450/2022.0222-22. Epub 2022 Nov 25. PMID 36580029
- [Derived] Pierelli L, De Rosa A, Falco M, Papi E, Rondinelli MB, Turani F, Weltert L. Preoperative Sucrosomial Iron Supplementation Increases Haemoglobin and Reduces Transfusion Requirements in Elective Heart Surgery Patients: A Prospective Randomized Study. Surg Technol Int. 2021 Oct 28;39:321-328. doi: 10.52198/21.STI.39.CV1512. PMID 34710946